CLINICAL TRIAL: NCT02967718
Title: Clinical Observation of CHD Phlegm and Blood-stasis Syndrome Patients
Brief Title: Innovation Research of Differentiation and Treatment Methods Based on CHD Phlegm and Blood Stasis Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jingqing Hu (Other)
Responsible Party: Sponsor-Investigator, Jingqing Hu, Director of Institute of Basic Theory of Traditional Chinese Medicine, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: 2014CB542903
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Control group: the healthy patients
- Metabolic syndrome group: Include patients who are accordance with diagnostic criteria of metabolic syndrome
- CHD stable stage group: Include patients who are accordance with diagnostic criteria of asymptomatic angina, stable angina or stable (more than 1 month) acute coronary syndrome
- Acute coronary syndrome group: Include patients who are accordance with diagnostic criteria of unstable angina or non-ST-segment elevated myocardial infarction
- PCI or CABG group: Include the patients who will undergo percutaneous coronary intervention of coronary artery bypass grafting
- CHD heart failure group: Include the patients who suffered heart failure cause by CHD

SUMMARY:
Coronary heart disease is still the major cause of death in China. Chinese medicine plays more and more important role in CHD prevention and treatment. Phlegm and blood stasis are its major pathological basis. Based on that, the investigator aims to evaluate the evolutionary process of CHD phlegm-blood stasis syndrome by large samples, multi-centre, cross-section observation combining with longitudinal tracking on-site survey method so as to guide the clinical treatment of CHD.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is a major cause of myocardial infarct (MI) and death induced by atherosclerosis or coronary artery spasm. Despite improvements in interventional and pharmacological therapy for acute MI, the mortality early after AMI remains high. Nowadays, as our life quality develops and dietary structure changes, the morbidity of hyperlipidemia dramatically increased. Based on the Chinese medicine, hyperlipidemia belongs to phlegm and it's the basis of atherosclerosis, blood-stasis is the pathological basis of ischemia. Therefore, the investigator proposes that phlegm and blood-stasis syndrome is the main differentiation on CHD. Based on that, the investigator prospectively and retrospectively explores the evolutionary process of CHD phlegm-blood stasis syndrome by large samples, multi-centre, cross-section observation combining with longitudinal tracking on-site survey method.It will provide evidence and guidance to the future clinical treatment using Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or metabolism syndrome people
* Clinical diagnosis of CHD stable stage or acute coronary disease or CHD heart failure

Exclusion Criteria:

* Any inflammation, fever, trauma, burn or operation within 1 week
* Obstructive pulmonary disease
* Cerebral vascular disease
* Severe renal or hepatic dysfunction
* Malignant neoplasms
* Hematopoietic system disease
* Sever mental disease

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, metabolic or coronary heart disease people, whose age is between 35-85 years old, either female or male, without any inflammation, fever, trauma, burn or operation within 1 week.
Sampling Method: Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Integrative Hospital of Beijing, Beijin, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang J, Tong H, Jiang L, Hu J. Dietary Patterns Associated With Heat Retention in Blood Vessel Syndrome (HRBVS) in Coronary Heart Disease: A Cross-Sectional Study. Int J Gen Med. 2025 Mar 5;18:1283-1294. doi: 10.2147/IJGM.S510507. eCollection 2025. PMID 40062358